CLINICAL TRIAL: NCT04884841
Title: Development and Validation of Models to Predict Postoperative Complications for Patients With Cardiac Surgery
Acronym: DV_model_CS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Yuefu Wang, Principal Investigator, Clinical Professor, China National Center for Cardiovascular Diseases
Other Study IDs: Prediction Model of CS
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with postoperative complications: Patients with postoperative complications
  Interventions: Other: Patients diagnosed with postoperative complications
- Patients without postoperative complications: Patients without postoperative complications
  Interventions: Other: Patients without postoperative complications

INTERVENTIONS:
Other: Patients diagnosed with postoperative complications — Patients diagnosed with postoperative complications (Acute kidney injury, Chronic Kidney disease, Infection, Delirium, MACCE, Myocardial infarction, Postoperative pulmonary complications, major bleeding, ECMO, IABP....)
  Groups: Patients with postoperative complications
Other: Patients without postoperative complications — Patients without postoperative complications
  Groups: Patients without postoperative complications

SUMMARY:
Patients undergoing cardiac surgery is routinely performed in clinical scenarios, highly postoperative morbidities and long-term mortality should be modified. A simple risk prediction model incorporating risk factors can help guide clinical decision making, patient counseling and treatment planning.

DETAILED DESCRIPTION:
Patients undergoing cardiac surgery is routinely performed in clinical scenarios, highly postoperative morbidities and long-term mortality should be modified.A nomogram is a pictorial representation of a scoring model that possesses a simple user interface and shows favorable predictive performance. By integrating a patient's diverse determinant variables, a nomogram can provide a personalized probability for quantitative predictions of the incidence of an outcome of interest.Therefore, we conducted a retrospective study to assess the incidence, risk factors and outcomes associated with major complications patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

Age more than 18 years Undergoing Cardiovascular surgery

Exclusion Criteria:

Missing primary outcomes or variables

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who are going to have an cardiovascular operation.
Sampling Method: Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
postoperative complications: acute kidney injury | 30 dyas
  Diagnosed acute kidney injury (KDIGO)
postoperative complications: Chronic Kidney disease | 30 days, as follow up
  Diagnosed Chronic Kidney disease
postoperative complications: Infection | 30 days
  Diagnosed infection
postoperative complications: delirium | 30 days
  Diagnosed delirium (CAM,CAM-ICU)
postoperative complications: MACCE | 30 days, as follow up
  Diagnosed MACCE
postoperative complications: major bleeding | 30 days
  Diagnosed major bleeding
postoperative complications: postoperative pulmonary complications | 30 days
  Diagnosed postoperative pulmonary complications
postoperative complications: ECMO | 30 days
  patients with ECMO
postoperative complications: IABP | 30 days
  patients with IABP
Ventilation time | Through study completion, an average of 7 days
  Number of hours the patient with mechanical ventilation
Length of ICU stay | Through study completion, an average of 30 days
  Number of days the patient stays in the intensive care unit

SECONDARY OUTCOMES:
Total hospital costs | Through study completion, an average of 30 days
  Total cost of the stay in the hospitalization (USD)
ICU costs | Through study completion, an average of 30 days
  Total cost of the stay in the intensive care unit (USD)
Length of hospital stay | Through study completion, an average of 30 days
  Number of days the patient stays in the hospital
Length of postoperative hospital stay | Through study completion, an average of 30 days
  Number of days the patient stays in the hospital after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yuefu Wang, MD, Principal Investigator — China National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, China National Center for Cardiovascular Diseases, CAMS&PUMC, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided